CLINICAL TRIAL: NCT06183450
Title: Hearing and Cognition in Aging Adults
Acronym: ACAV
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/22/0252; 2023-A01415-40 (Other: ID-RCB)
Record Dates: First submitted 2023-12-06; First posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Presbycusis
Keywords: presbycusis; aging; cognitive decline; speech in noise; sound localisation; hearing loss
MeSH Terms: conditions — Presbycusis; Cognitive Dysfunction; Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hearing subject: Adult normal hearing subjects, evaluated annually for 5 years,
  Interventions: Diagnostic Test: auditory level; Diagnostic Test: cognitive level; Diagnostic Test: quality of life level

INTERVENTIONS:
Diagnostic Test: auditory level — * Evaluation of auditory thresholds through audiometric tests.
  * Evaluation of speech comprehension in noise through a vocal audiometry test in noise (FraMatrix).
  * Evaluation of spatial auditory behavior and spatial precision using a spatial discrimination test (Minimum Audible Angle) and a static sound localization test in virtual reality.
Diagnostic Test: cognitive level — * Evaluation of attention and short-term memory functions with verbal and non-verbal tasks: Digit Span Test and Reading Span Test.
  * Evaluation of inhibition capacities using the Stroop Test.
  * Evaluation of executive functions, visual attention, reasoning, and mental arithmetic using the Raven's Matrix test.
Diagnostic Test: quality of life level — - Evaluation of quality of live level via Speech, Spatial and Qualities of Hearing Scale (SSQ-12) and EuroQol-5D questionnaires.

SUMMARY:
This cohort study is expected to provide valuable insights into the complex interplay between auditory and cognitive functions and how they change over time. The results of this study will have important implications for the prevention, diagnosis, and treatment of age-related hearing and cognitive disorders

DETAILED DESCRIPTION:
The aim of the study is to identify the early perceptual and cognitive alterations related to age-related hearing loss or presbycusis, establish a correlation between the degree of hearing loss and the deterioration of cognitive functions, and examine the effectiveness of hearing loss management in reversing observed cognitive impairments. This project has the potential to shed light on the importance of early detection of hearing impairments in preventing cognitive decline. The data collected from this cohort, rigorously assessed for both auditory and cognitive functions, could serve as the basis for several high-level scientific investigations.

ELIGIBILITY:
Inclusion Criteria:

* Normal hearing (Pure Tone Audiometry < or = 20 dB)
* Residency in one of the three neighborhoods :
* Affiliation with a social security system

Exclusion Criteria:

* Individuals under guardianship, trusteeship or curators
* History of neurological pathologies
* Taking of psychotropic medication.

Ages: 45 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adult normal hearing subjects aged between 45 and 50 years old.
Sampling Method: Probability Sample
Enrollment: 262 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2033-01 (Estimated); Study Completion 2033-01 (Estimated)

PRIMARY OUTCOMES:
Pure-ton audiometry | 5 years
  Pure-tone audiometry will be evaluated by collecting the threshold in air and bone conduction for both ears on each frequency tested (125-250-500-1000-2000-4000 and 8000 Hz), as well as the average hearing loss (MAP ) on all five frequencies.

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu Marx, Pr, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Ecole d'audioprothèse, Cahors, France

IPD SHARING:
Plan to Share IPD: No